CLINICAL TRIAL: NCT00517361
Title: A Phase II Study of Carboplatin and Bevacizumab (Avastin) Combination Therapy for ER Negative, PR Negative, and HER2/Neu Negative Metastatic Breast Cancer
Brief Title: Phase II Study of Carboplatin and Bevacizumab (Avastin) for ER Neg, PR Neg, and HER2/Neu Neg Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has been terminated due to poor accrual
Sponsor: University of Chicago (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15578A
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Results first posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-03

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carboplatin + Avastin (Experimental)
  Interventions: Drug: carboplatin; Drug: bevacizumab

INTERVENTIONS:
Drug: carboplatin — AUC 6 in 250mL saline IV over 30 minutes
Drug: bevacizumab — 15mg/kg in 100mL saline IV over 60 - 90 minutes
  Other Names: Avastin

SUMMARY:
The purpose of this study is to determine the progression free survival (PFS) of metastatic ER, PR and HER2/neu negative breast cancers to the combination of carboplatin and bevacizumab (Avastin®) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed ER, PR and HER2/neu negative (FISH ratio of <2.0 or IHC <1+) metastatic breast cancer. Locally advanced or recurrent disease is also eligible.
* Patients must have measurable disease
* Patients must not have received prior chemotherapy for metastatic breast cancer (not including adjuvant therapy). Patients should be > 4 weeks from their most recent chemotherapy or radiation therapy treatment.
* Age >18 years
* ECOG performance status <1 (Karnofsky >80%).
* Patients must have normal organ and marrow function as defined below:
* absolute neutrophil count >1,500/uL
* platelets >100,000/uL
* total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) <2.5X institutional upper limit of normal
* creatinine within normal institutional limits OR creatinine clearance>60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* PT INR < 1.5 (Unless patient is on anticoagulation)
* urine protein <1+
* Tissue from the primary tumor must be available for correlative studies
* Women of child-bearing potential must agree to use adequate contraception
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had prior therapy with platinum agents or a VEGF inhibitor are not eligible.
* Patients may not be receiving any other investigational agents.
* Patients with known brain metastases will be excluded
* Patients may have had prior radiation therapy, provided the patient has measurable disease and there has been clear progression since the completion of radiation therapy. Patients who have had radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to therapy administered more than 4 weeks earlier will be excluded.
* Patients with significant cardiac dysfunction will be excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study, breastfeeding should be discontinued.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with carboplatin or the other agents administered during the study.
* Patients with evidence of bleeding diathesis or coagulopathy.
* Patients with inadequately controlled hypertension will be excluded
* Patients who have had a stroke or TIA within 6 months of registration will be excluded.
* Patients with a history of hypertensive crisis or hypertensive encephalopathy will be excluded.
* Patients with a history of abdominal fistula, GI perforation, or intra-abdominal abscess within 6 months of registration.
* Patient with history of serious non-healing wound, ulcer or bone fracture.
* Patients with major surgery, open biopsy, or significant traumatic injury within 28 days of registration or anticipated need for surgery during course of study treatment.
* Patients with a history core biopsy or other minor surgery, excluding venous access device (VAD) placement, within 7 days of registration.
* Patients with active second malignancy.
* Known hypersensitivity to any component of bevacizumab (Avastin®).
* Peripheral neuropathy > Grade 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-08; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Nanda, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - Oncology Specialists, Park Ridge, Illinois

RESULTS

PARTICIPANT FLOW:
Groups:
- Carboplatin + Avastin: Carboplatin in 250mL saline IV over 30 minutes and Avastin (Bevacizumab) 15mg/kg in 100mL saline IV over 60 - 90 minutes
Period: Overall Study
Arm/Group | Carboplatin + Avastin
Started | 11
Completed | 0 (This study has been terminated due to poor accrual.)
Not Completed | 11
Not completed — Death | 6
Not completed — The study was terminated | 5

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin + Avastin
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression is defined using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(3):205-216, 2000], as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions, or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Up to 5 years
Population: This study has been terminated due to poor accrual.
Arm/Group | Carboplatin + Avastin
Number analyzed (Participants) | 0

2. Secondary Outcome: Response Rate
Description: Response is defined using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(3):205-216, 2000]: Complete Response (CR), Disappearance of all target lesions or disappearance of all non-target lesions and normalization of tumor marker level; Partial Response (PR), At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD since the treatment started, or persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits.
Time Frame: Up to 5 years
Population: This study has been terminated due to poor accrual.
Arm/Group | Carboplatin + Avastin
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response
Time Frame: Up to 5 years
Population: This study has been terminated due to poor accrual.
Arm/Group | Carboplatin + Avastin
Number analyzed (Participants) | 0

4. Secondary Outcome: Correlation of Response to BRCA1 Methylation Status
Description: The methylation status of the tumor is defined using Methylation Specific polymerase chain reaction and/or pyrosequencing.
Time Frame: Up to 5 years
Population: This study has been terminated due to poor accrual.
Arm/Group | Carboplatin + Avastin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Carboplatin + Avastin
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin + Avastin (N=11)
nausea (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
pain (General disorders) | 1 (1)
severe weakness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin + Avastin (N=11)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
pain (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Creatinine increased (Investigations) | 1 (1)
Ear, nose and throat examination abnormal (Investigations) | 1 (1)
Hemoglobin (Investigations) | 2 (2)
Hemoglobin decreased (Investigations) | 2 (2)
Hyperglycemia (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1)
Leukocytes (Investigations) | 3 (3)
Neutrophil count decreased (Investigations) | 2 (2)
Neutrophils (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 2 (2)
Platelets (Investigations) | 6 (6)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hemorrhage - Other (Specify) (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Vascular - Other (Specify) (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No